CLINICAL TRIAL: NCT03378505
Title: Living Purposefully: The Role of Mobile App JOOL in Promoting Well-being and Academic Success
Brief Title: Impact of Mobile App on Purpose and Well-Being Among College Students
Acronym: PWB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-1371; A271000 (Other: UW Madison); SOHE\CONSUMER SCIENCE\CONS SCI (Other: UW Madison)
Record Dates: First submitted 2017-12-04; First posted 2017-12-19 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Healthy
MeSH Terms: interventions — Microscopy, Interference

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two conditions. Half of the participants will be required to use a daily check-in mobile app that promotes alignment of daily behaviors with their individualized life purpose. The other half of participants will complete brief bi-weekly reflections. Alternative assignment provided for non-participating students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile App (Experimental): Half of the students randomly assigned
  Interventions: Behavioral: Mobile App
- Reflection (Experimental): Half of the students randomly assigned
  Interventions: Behavioral: Reflection

INTERVENTIONS:
Behavioral: Mobile App — Purposeful Living Mobile App JOOL to be used daily
  Other Names: JOOL
  Arms: Mobile App
Behavioral: Reflection — Bi-weekly online reflection question
  Arms: Reflection

SUMMARY:
This study will examine the impact of a mobile app (JOOL) focused on promoting purposeful living on student health behaviors, academic performance, self-regulation, well-being, resiliency, and self-efficacy.

DETAILED DESCRIPTION:
Participants will be recruited from a large undergraduate classroom. Participants will be randomly assigned to one of two conditions and asked to complete either online reflections or engage with a mobile app over the course of the semester. Students who elect to not participate will be provided an alternate assignment to complete, to be coordinated by their teaching assistant. Participants will additionally be asked to complete (1) a pre-survey, (2) post-survey, and follow-up survey 14 days after the class concludes. The study will examine changes in health-related behaviors, resiliency, well-being, and self-efficacy reported between the start and conclusion of semester/study.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Enrolled in Consuming Happiness course during the Spring 2017-18 semester.
* Must have access to WiFi, cellular service or computer with internet connection and web browser.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Health Behaviors | 14 weeks post start (1 semester)
  Expected increase in self-report of behaviors promoting academic achievement, physical health, well-being, and purpose from time of pre survey to post survey.
Change in Resiliency | 14 weeks post start (1 semester)
  Brief Resiliency Scale (BRS) used to measure resiliency, or ""the ability to bounce back or recover from stress" (Smith et al., 2008). 6 items using Likert scale strongly disagree (1) to strongly agree (5). Score will be summed for one total score and can range from 6 to 30, with 6 indicating low resilience and 30 indicating high resilience. No clinical cut off. Expected increase no change in scores from pre and post.
Change in Self-Regulation | 14 weeks post start (1 semester)
  Self-Regulation Scale (SRQ) short form used to measure self-regulation, or ""the ability to develop, implement, and flexibly maintain planned behavior in order to achieve one's goal" (Brown, Miller, & Lawendowski, 1999). 31 items using a Likert scale strongly disagree (1) to strongly agree (5), with 14 reverse coded. Scores will be summed for one total score ranging from 31 to 155. 31 indicates low self-regulation and 155 indicates high self-regulation. No clinical cut off. Expected increase or no change in scores from pre and post.
Change in belief of ability to perform difficult tasks or cope with diversity | 14 weeks post start (1 semester)
  Generalized Self-Efficacy Scale used to measure self-efficacy, or "the optimistic self-belief that one can perform novel or difficult tasks or cope with diversity" (Schwarzer, 1992). 10 items on a Likert scale from Not true at all (1) to Exactly true (4). Responses will be summed for one total score, ranging from 10 to 40. 10 indicates low self-efficacy, 40 indicates high self-efficacy. No clinical cut off. Expected increase or no change in scores from pre and post.
Change in Well-Being | 14 weeks post start (1 semester)
  The WHO (Five) Well-Being Index (WHO-5) measures well-being, defined as the subjective quality of life based on positive mood (good spirits, relaxation), vitality (being active and waking up fresh and rested), and general interest (being interested in things). 5 items on a Likert scale ranging from all of the time (5) to at no time (1). Responses will be summed for one total score ranging from 0 to 25. 0 indicates low well-being and 5 indicates high well-being. Score below 13 indicates poor well-being. Expected increase or no change in scores from pre and post.

SECONDARY OUTCOMES:
Change in Health Behaviors | 14 days (2 weeks) after end of study (16 weeks post start)
  Expected increase or no change in reported health behaviors around academic achievement and well-being from time of post survey. To be completed 2 weeks after post-survey.
App Perceptions | 14 days (2 weeks) after end of study (16 weeks post start)
  Feedback on perceptions of the mobile app and information on continued use behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- School of Human Ecology, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared with researchers not directly associated with the study and/or listed on the IRB.